CLINICAL TRIAL: NCT00368095
Title: The Rajavithi Prospective Cohort Study on Community's Member Health (HPH-cohort Study)
Brief Title: Rajavithi Health Promotion Project (Population Base Cohort)
Status: Active, not recruiting | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: RVH_CER_004
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus; Hypertension; Dyslipidemia; Obesity; Cardiovascular Disease; Coronary Artery Disease
Keywords: DM; HT; Dyslipidemia; Obesity; Cardiovascular disease; Cerebrovascular disease; Myocardial infarction; stroke; Metabolic syndrome; CVD-CAD
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias; Obesity; Cardiovascular Diseases; Coronary Artery Disease; Cerebrovascular Disorders; Myocardial Infarction; Stroke; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human Genetic Bank will be storaged in Biomolecular center Rajavithi Hospital for determine the gene that influence the specific disease in the population

INTERVENTIONS:
Behavioral: Intensive Education for Metabolic Syndrome Patients — Excercise, Intensive diatary program
  Other Names: Patient with Metabolic Syndrome will be advised fro improve health status and genetic test will be apply

SUMMARY:
Metabolic Syndrome (hypertension, diabetes mellitus, obesity, cerebrovascular-cardiovascular disease) In Community Survey was performed in central Bangkok.

Prospective Cohort and intensive educated intervention (health promotion program in specific high risk groups) were performed. The aim of the study is to identify high risk patients who can develop serious complications from metabolic syndrome. An analysis of health outcomes in multiple dimensions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or more
* Informed consent
* Living in selected community (Health Promotion area of Rajavithi Hospital)

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population in Dindang destrict Bangkok
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2006-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand; Piyathida Harnsomboonrana, M.D., Study Director — Department of Medical Services Ministry of Public Health of Thailand; Wilai Pauvilai, M.D., Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand